CLINICAL TRIAL: NCT02704455
Title: Registry Study on Primary Ciliary Dyskinesia in Chinese children-a Multicenter, Prospective Cohort Study
Brief Title: Registry Study on Primary Ciliary Dyskinesia in Chinese Children
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shengjing Hospital (Other); Capital Institute of Pediatrics, China (Other); Shanghai Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); The First Affiliated Hospital of Xiamen University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Other Study IDs: BCHlung005
Record Dates: First submitted 2016-03-03; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: children
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a multicenter, prospective cohort study of patients diagnosed with primary ciliary dyskinesia, the clinical information of recruited patients, including clinical manifestations, lung function, chest imaging, quality of life and other indicators, will be followed for 10 years.

DETAILED DESCRIPTION:
All new cases of primary ciliary dyskinesia which was confirmed or diagnosed at each center from the beginning of the study are made the investigation of the clinical manifestations and specific tests by the standard diagnostic process.Then all the patients' following clinical data will be followed for 10 years (once per six month): clinical manifestations, lung function, chest imaging (once per year), quality of life and other indicators.

ELIGIBILITY:
Inclusion Criteria: A included patient must be coincident with all the following items:

* Age 0~18 years old
* Any organ system symptoms consistent with PCD and being conform to the clinical diagnostic standard of Katergener syndrome or being coincident with at least two following specific tests:
* Abnormal ciliary beat frequency or movement by the high speed photography microscope
* Abnormal ciliary structure through the electronic microscopy
* The nasal NO decreased significantly
* The target gene mutation found
* The clinical diagnostic criteria of the Katergener syndrome: ① bronchial expansion; ② sinusitis or nasal polyps; ③ transposition of viscera and (or) dextrocardia.
* If all the typical clinical manifestations but only 1 specific test with positive results, can also be included in the registration of suspected PCD cases
* Consent to provide the related clinical specimen to the certain hospital
* The guardians of the patients fully understand the purpose of the study, volunteer their children to participate in this study, and sign informed consent.

Exclusion Criteria: Subject will be excluded if she or he has one of the following:

* It is unable to provide complete medical records or the current condition can not accept the diagnosis process
* She or he cannot agree to participate in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as primary ciliary dyskinesia at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2030-05 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung function on the spirometry | 10 years
  forced expiratory volume at one second (FEV1) in Liter

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China;China National Clinical Research Center for Respiratory Diseases; Baoping Xu, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China;China National Clinical Research Center for Respiratory Diseases

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Liu Y, Wang L, Tian X, Xu KF, Xu W, Li X, Yue C, Zhang P, Xiao Y, Zhang X. Characterization of gene mutations and phenotypes of cystic fibrosis in Chinese patients. Respirology. 2015 Feb;20(2):312-8. doi: 10.1111/resp.12452. Epub 2015 Jan 8. PMID 25580864
- [Background] Hogg C, Bush A. Genotyping in primary ciliary dyskinesia: ready for prime time, or a fringe benefit? Thorax. 2012 May;67(5):377-8. doi: 10.1136/thoraxjnl-2011-201320. Epub 2012 Jan 9. No abstract available. PMID 22232363
- [Background] Shapiro AJ, Zariwala MA, Ferkol T, Davis SD, Sagel SD, Dell SD, Rosenfeld M, Olivier KN, Milla C, Daniel SJ, Kimple AJ, Manion M, Knowles MR, Leigh MW; Genetic Disorders of Mucociliary Clearance Consortium. Diagnosis, monitoring, and treatment of primary ciliary dyskinesia: PCD foundation consensus recommendations based on state of the art review. Pediatr Pulmonol. 2016 Feb;51(2):115-32. doi: 10.1002/ppul.23304. Epub 2015 Sep 29. PMID 26418604
- [Background] Noone PG, Leigh MW, Sannuti A, Minnix SL, Carson JL, Hazucha M, Zariwala MA, Knowles MR. Primary ciliary dyskinesia: diagnostic and phenotypic features. Am J Respir Crit Care Med. 2004 Feb 15;169(4):459-67. doi: 10.1164/rccm.200303-365OC. Epub 2003 Dec 4. PMID 14656747